CLINICAL TRIAL: NCT05433519
Title: Z 32104 - Diagnostic Accuracy of a Novel Machine Learning Algorithm to Estimate Gestational Age
Brief Title: Diagnostic Accuracy of a Novel Machine Learning Algorithm to Estimate Gestational Age
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 21-3115
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-12

CONDITIONS: Gestational Age; Machine Learning; Pregnancy Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum, and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant Women: Pregnant women with gestational age established at less than 14 weeks of gestation

SUMMARY:
This is a prospective cohort study of women enrolled early in pregnancy, with randomization to determine the timing of three follow-up visits in the second and third trimester. At each of these follow-up visits, investigators will assess gestational age with the FAMLI technology and compare that estimate to the known gestational age established early in pregnancy.

DETAILED DESCRIPTION:
The primary purpose of this research is to assess the diagnostic accuracy of the FAMLI Technology, a novel machine learning-based tool for gestational age assessment that can run on a smart phone or tablet. Study staff will enroll 400 pregnant volunteers prior to 14 completed gestational weeks and obtain accurate "ground truth" gestational age dating with standard ultrasound biometry, using the crown-rump length. These participants will then be asked to return for three follow-up visits, which will include a routine sonogram performed by a trained sonographer and the collection of a set of blind sweep cineloop videos using a low-cost, battery-operated device. The research will be conducted in Chapel Hill, North Carolina (at the University of North Carolina Hospital and/or sites associated with UNC OBGYN) and in Lusaka, Zambia (at the University Teaching Hospital or Kamwala District Health Centre). Approximately equal numbers of participants will be enrolled from each country.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* viable intrauterine pregnancy at less than 14 0/7 weeks of gestation
* ability and willingness to provide written informed consent
* intent to remain in current geographical area of residence for the duration of study
* willingness to adhere to study procedures

Exclusion criteria:

* maternal body mass index = 40 kg/m^2
* multiple gestation (i.e., twins or higher order)
* major fetal malformation or anomaly
* any other condition (social or medical) that, in the opinion of the study staff, would make study participation unsafe or complicate data interpretation.

Ages: 18 Years to 59 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women at 14 weeks or earlier gestation
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of FAMLI Technology | From 14 through 27 completed weeks of gestation
  Difference in mean absolute error (MAE) of the index test and clinical reference standard in the primary evaluation window

SECONDARY OUTCOMES:
Mean absolute error in the secondary evaluation window | From 28 through 36 completed weeks of gestation
  Difference in mean absolute error (MAE) of the index test and clinical reference standard in the secondary evaluation window

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Stringer, MD, Principal Investigator — University of North Carolina
Locations (2):
- University of North Carolina, Chapel Hill, North Carolina, United States
- University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: 9-36 months following publication
Access Criteria: noted above

REFERENCES:
- [Derived] Stringer JSA, Pokaprakarn T, Prieto JC, Vwalika B, Chari SV, Sindano N, Freeman BL, Sikapande B, Davis NM, Sebastiao YV, Mandona NM, Stringer EM, Benabdelkader C, Mungole M, Kapilya FM, Almnini N, Diaz AN, Fecteau BA, Kosorok MR, Cole SR, Kasaro MP. Diagnostic Accuracy of an Integrated AI Tool to Estimate Gestational Age From Blind Ultrasound Sweeps. JAMA. 2024 Aug 27;332(8):649-657. doi: 10.1001/jama.2024.10770. PMID 39088200

DOCUMENTS (2):
  • Study Protocol (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT05433519/Prot_002.pdf
  • Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT05433519/SAP_001.pdf